CLINICAL TRIAL: NCT07270978
Title: Phase Ib Study of Anti-CD3 x Anti-CD33 Bispecific Antibody (CD33Bi) Armed Fresh Peripheral Blood Mononuclear Cells (CD33 FPBMC) in Patients With Measurable Residual Disease (MRD)+ Acute Myeloid Leukemia or Myelodysplastic Syndrome
Brief Title: Phase Ib Study of CD33 FPBMC in Patients With MRD+ AML or MDS
Acronym: AML-MDS 001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Daniel R. Reed, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 302332
Record Dates: First submitted 2025-11-17; First posted 2025-12-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD33 FPBMC + hypomethylating agent with or without venetoclax (Experimental): 4 weekly infusions of CD33 fresh peripheral blood mononuclear cells (FPBMC) followed by 4-6 weeks of hypomethylating agent with/without venetoclax.
  Interventions: Drug: CD33 FPBMC

INTERVENTIONS:
Drug: CD33 FPBMC — Participants will receive up to 4 cycles of 4 weekly infusions of CD33 infusions followed by 4-6 weeks of a hypomethylating agent with or without venetoclax according to standard clinical care.

SUMMARY:
The purpose of this study is to understand the safety and estimate the efficacy of combining anti-CD3 x anti-CD33 bispecific antibody (CD33Bi) armed fresh peripheral blood mononuclear cells (CD33Bi FPBMC) for patients with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) where they still have detectable disease ("MRD+") after some treatment. Participants receive 4 weekly doses of CD33 FPBMC by intravenous infusion followed by 4-6 weeks of standard treatment with a hypomethylating agent (type of treatment such as decitabine or azacitidine) and possibly a drug called venetoclax. This is considered 1 cycle of study treatment and may be repeated up to 4 times during the study.

DETAILED DESCRIPTION:
Once subjects are determined to be eligible, white blood cells (lymphocytes) are collected via leukapheresis procedure. The T cells in the mononuclear cells are coated with bispecific antibody to activate the T cells and the mononuclear cells are reinfused into the patients so the T cells can multiply and kill AML/MDS cells.

At least 72 hours after the leukapheresis procedure, study treatment will start. Participants receive 4 weekly doses of CD33 FPBMC by intravenous infusion followed by 4-6 weeks of standard treatment with a hypomethylating agent (type of treatment such as decitabine or azacitidine) and possibly a drug called venetoclax. This is considered 1 cycle of study treatment and may be repeated up to 4 times during the study.

After about 2 cycles of study treatment, participants will have another leukapheresis procedure. Before, throughout and following study treatment, research blood will be collected to better understand immune response. Disease status will be checked regularly during and after study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults: ≥18 years of age
2. Diagnosis of either:

   1. Newly diagnosed or relapsed/refractory AML who have received at least 2 cycles of azacitidine and venetoclax
   2. Relapsed/ refractory (R/R) MDS who have received at least 2 prior cycles of azacitidine and venetoclax or single agent hypomethylating agent for at least 4 cycles
   3. Relapsed/refractory (R/R) MDS/MPN overlap syndromes like CMML who have received at least 2 prior cycles of azacitidine and venetoclax or single agent hypomethylating agent for at least 4 cycles
3. For patients with targetable mutations (IDH1, IDH2, KMT2A, or FLT3): Receipt of and/or decision not to receive associated inhibitor.
4. Patients with R/R MDS or R/R MDS/MPN overlap syndromes must have at least one of the following:

1) Bone marrow blasts >5% and higher than previous evaluation by at least 5% 2) Progression to AML (≥20% blasts) 3) Appearance of previously absent leukemic blasts in peripheral blood 4) Absolute neutrophil count <1 x 109/L and 50% below best unsupported on-study value 5) Platelet count <100 x 109/L and 50% below best unsupported on-study value 6) Hemoglobin <11g/dL, and ≥2 g/dL reduction from best unsupported on-study value 7) Increase of the volume of transfused red blood cells by more than 30% in an 8-week period 8) Increase of the number of transfused platelet units by more than 30% in an 8-week period In the case of criteria 4-8 above, no reasonable alternative explanation such as drug toxicity should be identified.

5. Patients with AML must have:

1. Persistent or recurrent MRD positivity defined by presence of blasts ≥5% and <20% AND/OR disease detected by multiparametric flow cytometry (MFC) at a level of ≥0.1%, AND/OR persistent genomic mutations other than those found most with CHIP (DNMT3A, ASXL1, TET2) AND/OR persistent cytogenetic abnormalities related to underlying myeloid neoplasm
2. Residual blasts must be positive for CD33 expression at any level
3. Myeloblasts must be <20%

   6. Left Ventricular Ejection Fraction (LVEF) ≥ 45% at rest (MUGA or echocardiogram)

   7. Performance status ≤ 2 (ECOG Scale)

   8. Females of childbearing potential and males must agree to use an effective method for contraception for the duration of the treatment with study drug plus 90 days (duration of sperm turnover). Males must also abstain from sperm donations during study treatment and for at least 90 days after the last dose of study drug.

   9. Ability to provide informed consent and provision of written informed consent In order to be eligible to participate in the dose expansion portion of this study, an individual must meet all criteria that apply to the R/R MDS or R/R AML population (Newly diagnosed patients and patients with MDS/MPN overlap syndromes are not eligible for the expansion phase of the study).

In order to be eligible to participate in the dose expansion portion of this study, an individual must meet all criteria that apply to the R/R MDS or R/R AML population (Newly diagnosed patients and patients with MDS/MPN overlap syndromes are not eligible for the expansion phase of the study).

Exclusion Criteria:

1. Pregnancy or lactation
2. Prior treatment with anti-CD33 therapy
3. Patients who are being actively considered for stem cell transplant. This does not exclude patients that may be eligible for stem cell transplant at some future (undetermined) date.
4. Clinically significant organ dysfunction, defined as any of the following:

   * AST or ALT >3x the upper limit of normal (ULN)
   * Total bilirubin >1.5x the ULN, unless due to ongoing hemolysis or Gilbert's syndrome, in which case > 3.0 mg/dL
   * Absolute lymphocyte count (ALC) < 300 lymphocytes/microliter
   * Creatinine clearance <30 mL/min
   * Active serious infection not controlled by oral or intravenous antibiotics (e.g. persistent fever or lack of clinical improvement despite antimicrobial treatment).
5. Patients that are platelet refractory with a platelet level of <30,000 platelets/microliter
6. Known human immunodeficiency virus (HIV) with detectable viral load.
7. Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection

   a. Note: Patients who have isolated positive hepatitis B core antibody (ie, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.
8. Patients with a prior or concurrent malignancy whose natural history or treatment is anticipated to interfere with the safety or efficacy assessment of the investigational regimen (according to the treating investigator).
9. Treatment with any antileukemic agents or chemotherapy (other than hypomethylating agents or venetoclax) agents in the last 7 days or 5 half-lives (whichever is sooner) before study entry.
10. Known allergy to hypomethylating agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
DLTs | From start of treatment through 7 days after the 4th infusion (for each participant)
  Escalation phase participants only

SECONDARY OUTCOMES:
Overall response rate (ORR) | During study treatment and for up to 3 years following intervention
  Based on MRD status (AML cohort) and IWG criteria1 (MDS cohort)
Disease status | During study treatment and for up to 3 years following intervention
  According to European LeukemiaNet (ELN) criteria (AML cohort) or IWG criteria (MDS cohort)
Progression free survival (PFS) | From baseline to disease progression or death from any cause, whichever comes first, assessed up to 3 yrs after last study drug administration
  European LeukemiaNet (ELN) criteria (AML cohort) or IWG criteria (MDS cohort)
Adverse Events (AEs) | During and up to 30 days after last study treatment (all reportable AEs) and during long term follow-up (up to 3 years) for serious AEs considered related to study treatment
  According to CTCAE v5

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Reed, MD, Principal Investigator — Assistant Professor; Lawrence Lum, MD, DSc, Study Director — IND Sponsor
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No